CLINICAL TRIAL: NCT04776785
Title: Effect of Self-Assembling Peptides on the Progression of Non-Cavitated Proximal Caries: A Randomized Controlled Clinical Trial
Brief Title: Effect of Self-Assembling Peptides on the Progression of Non-Cavitated Proximal Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Merve AKCAY, Assoc. Prof. Dr., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-TDU-DİŞF-0001
Record Dates: First submitted 2021-02-27; First posted 2021-03-02 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Proximal Caries
Keywords: Proximal caries, P11-4, CPP-ACFP, fluoride varnish

STUDY DESIGN:
Intervention Model Description: randomized controlled, three-arm parallel, double-blinded, split-mouth clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization was performed by a computer-generated random sorting sequence (sealed in opaque envelopes that sequentially numbered randomly selected through).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): In Group 1, one lesion will be received self-assembling peptide P11-4 solution (Curodont™ Repair, Credentis AG, Windisch, Switzerland) followed by 5% NaF varnish (Profluorid® Varnish, VOCO GmbH, Cuxhaven, Germany) (test 1). The other lesion will be received 5% NaF varnish alone (Profluorid® Varnish, VOCO GmbH, Cuxhaven, Germany) (control).
  At the 6th and 12th months after the clinical applications, Profluorid® Varnish application will be repeated for test 1 and control lesions.
  Interventions: Device: Curodont™ Repair; Device: Profluorid® Varnish
- Group 2 (Experimental): In Group 2, one lesion will be received self-assembling peptide P11-4 solution (Curodont™ Repair, Credentis AG, Windisch, Switzerland) followed by 5% NaF varnish (Profluorid® Varnish, VOCO GmbH, Cuxhaven, Germany) (test 1). The other lesion will be received CPP-ACP varnish containing 5% NaF (MI Varnish™, GC America Inc., Alsip, IL, USA) (test 2).
  At the 6th and 12th months after the clinical applications; Profluorid® Varnish application will be repeated for test 1 lesions, and MI Varnish™ application will be repeated for test 2 lesions.
  Interventions: Device: Curodont™ Repair; Device: MI Varnish™; Device: Profluorid® Varnish
- Group 3 (Active Comparator): In Group 3, one lesion will be received CPP-ACP varnish containing 5% NaF (MI Varnish™, GC America Inc., Alsip, IL, USA) (test 2). The other lesion will be received 5% NaF varnish alone (Profluorid® Varnish, VOCO GmbH, Cuxhaven, Germany) (control).
  At the 6th and 12th months after the clinical applications; MI Varnish™ application will be repeated for test 2 lesions, and Profluorid® Varnish application will be repeated for control lesions.
  Interventions: Device: MI Varnish™; Device: Profluorid® Varnish

INTERVENTIONS:
Device: Curodont™ Repair — It is a product used in biomimetic remineralization of initial carious lesions. The product consists of "smart" P11-4 peptide molecules (CUROLOX® TECHNOLOGY) that within the lesion the molecules self-assemble to a 3D matrix. This bio-matrix enables the regeneration of the tooth tissue.
  Test 1 lesions will be cleaned with a prophylaxis paste and isolated with cotton rolls. Then, the pellicle will be removed using 2% sodium hypochlorite (20 sec) and the inorganic deposits will be removed using 35% phosphoric acid (20 sec). The tooth surface will be rinsed with water and dried. Thereafter, Curodont™ Repair will be applied in compliance with the manufacturers' instructions and left for 5 minutes.
  Other Names: CURODONT™ REPAIR, Credentis AG, Windisch, Switzerland
  Arms: Group 1; Group 2
Device: MI Varnish™ — MI Varnish™ is a 5% sodium fluoride (NaF) varnish that has a desensitizing action when applied to tooth surfaces. The product also contains RECALDENT™ (CPP-ACP): Casein Phosphopeptide-Amorphous Calcium Phosphate. The application leaves a film of varnish on tooth surfaces and also facilitates the tooth remineralization.
  Test 2 lesions will be isolated with cotton rolls. Then, MI Varnish ™ will be applied as a thin layer in equal thickness with a disposable brush in accordance with the manufacturers' instructions. Thereafter, the tooth surface will be moistened with water or saliva to ensure that the material adheres to the applied area.
  Other Names: MI Varnish™, GC America Inc., Alsip, IL, USA
  Arms: Group 2; Group 3
Device: Profluorid® Varnish — Profluorid® Varnish is a 5% sodium fluoride (NaF) varnish for surface application to enamel and dentin. The product will adhere to wet surfaces and is tolerant to moisture and saliva. Profluorid® Varnish is an ethanolic suspension of colophony with artificial flavors and sweetened with xylitol. It is also used in the remineralization of initial caries.
  Control lesions will be isolated with cotton rolls. Then, Profluorid® Varnish will be applied as a thin layer in equal thickness with a disposable brush in accordance with the manufacturers' instructions. Thereafter, the tooth surface will be moistened with water or saliva to ensure that the material adheres to the applied area.
  Other Names: VOCO Profluorid® Varnish, VOCO GmbH, Cuxhaven, Germany

SUMMARY:
The aim of this randomized controlled, double-blinded, split-mouth clinical trial was to evaluate the efficacy of self-assembling peptide P11-4 solution (Curodont™ Repair) with fluoride varnish on the progression of non-cavitated proximal caries compared to casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) with fluoride varnish (MI Varnish™) sodium fluoride (NaF) varnish (Profluorid® Varnish).

The study included 300 permanent molars belonging to 150 children, aged between 7 to 13 years old, who had two non-cavitated proximal carious lesions.

DETAILED DESCRIPTION:
First, the subjects were randomly allocated to three main groups with 50 individuals in each. Then the carious lesions belonging to each subject were randomly assigned to two subgroups based on different treatment agents used: Group 1; P11-4+NaF/NaF, Group 2; P11-4+NaF/CPP-ACP+NaF, Group 3; CPP-ACP+NaF/NaF. Accordingly, test 1 lesions received P11-4+NaF combination, test 2 lesions received CPP-ACP+NaF varnish, and control lesions received NaF varnish alone. At the 6th and 12th months after the clinical applications, Profluorid® Varnish application was repeated for test 1 and control lesions, and MI Varnish™ application was repeated for test 2 lesions. At the end of the 12 months, carious lesion progression status was evaluated radiographically, by using independent visual reading, pair-wise visual reading, and digital subtraction radiography (DSR) methods.

ELIGIBILITY:
Inclusion Criteria:

* Children who had two permanent molars with non-cavitated proximal carious lesions that included one in the right jaw and the other one in the left jaw, and in contact with neighboring teeth,
* Non-cavitated proximal carious lesions which is radiographically extending into either the outer half of the enamel (E1), the inner half of the enamel (E2) or the outer third of the dentin (D1),
* Children who had not any systemic disease that prevents the application,
* Cooperative children who allowed to radiographic examinations and clinical applications.

Exclusion Criteria:

* There is caries/restoration on the different surface of the tooth to be treated,
* There is caries/restoration on the contact surface of the tooth adjacent to the tooth to be treated,
* Non-cavitated proximal carious lesions which is radiographically extending into the middle third of the dentin (D2) or the inner third of the dentin (D3),
* There is cavitation on the proximal surface of the tooth to be treated,
* Non-cooperative children who had not allow to radiographic examinations and clinical applications,
* Children and parents who denied the participation in the follow-up appointments.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
The assessment of lesion progression by digital subtraction radiography (DSR) | 12 months after the clinical applications
  The primary outcome of the study was assessment of lesion progression (change in the lesions' opacity) by DSR readings, at 12th month.

SECONDARY OUTCOMES:
The assessment of lesion progression by pair-wise visual reading of radiographs | 12 months after the clinical applications
  One of the secondary outcomes of the study was assessment of lesion progression (change in the lesions' opacity) assessed by pair-wise visual readings, at 12th month.
The assessment of lesion progression by independent visual reading of radiographs | 12 months after the clinical applications
  The other one of the secondary outcomes of the study was assessment lesion progression (change in the classification of the lesions' size with respect to E0-E2, D1-D3 radiographic scoring system) assessed by independent visual readings, at 12th month.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Akcay, assoc. prof., Study Chair — Izmir Katip Celebi Uni
Locations (2):
- Turkey (Türkiye) (2):
  - Izmir Katip Celebi Uni., Izmir
  - Izmir Katip Celebi University, Izmir